CLINICAL TRIAL: NCT01049828
Title: Resting-State Neural Connectivity in Patients With Subjective Tinnitus Without Bother
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: WU625296
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: Tinnitus
Keywords: Tinnitus; fcMRI; Neural Connectivity; Bother
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Slightly or Non-Bothered Tinnitus Group: Identified by a Tinnitus Handicap Index <36 and a subjective description of their tinnitus as no or slight "bother."
  A control group has been collected through a different study, i.e. no controls will be recruited in this study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No treatment for tinnitus will occur in this study.

SUMMARY:
Tinnitus is the occurrence of an auditory sensation without the presence of an acoustic stimulus. Approximately, 50 million people in the United States experience chronic tinnitus and 15 million of these people have bothersome tinnitus. Several studies have shown that people who are bothered by their tinnitus have difficulty in concentration and focus. Through imaging modalities we have deranged neural networks responsible for attention. Only 20 percent of patients diagnosed with tinnitus are severely bothered. We seek the following:

1. Match a group of non-bothered tinnitus patients on age and hearing status to an existing cohort of bothered tinnitus patients.
2. Assess the resting-state neural connectivity in patients with non-bothersome tinnitus. Findings from the comparison of functional connectivity magnetic resonance imaging (fcMRI) from subjects with bothersome tinnitus in our current rTMS clinical trial to normal age-matched controls without tinnitus demonstrates that subjects with bothersome tinnitus have dramatic alterations in cortical attention and control networks. Our hypothesis is that the fcMRI-defined changes in the attention and control networks reflect the impact of excessive auditory stimulation in patients with bothersome tinnitus and explains the difficulty with concentration, short-term memory, and other common problems. To fully test this hypothesis we need to obtain fcMRI of the attention network among subjects with tinnitus but without bother and compare the status of their neural networks with those of tinnitus subjects with bother and with normal controls.
3. Compare the resting cortical networks in subjects with non-bothersome tinnitus to subjects with bothersome tinnitus and subjects without tinnitus Our null hypothesis is that there are no differences in the resting-state cortical networks, especially the attention and control networks, between tinnitus patients who do not experience bother, tinnitus patients who do experience bother, and subjects without tinnitus. Through fcMRI, we will examine correlations in blood oxygen level dependent (BOLD) signals in established auditory, attention, control, and other brain regions in the resting brain and compare these findings to already collected fcMRI scans of bothered tinnitus patients, and controls (patients without tinnitus).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 45 and 60 years
* Subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or greater
* A recent audiogram (within 6 months)
* Either "not bothered" or "bothered a little" on the Global Bothersome scale
* Able to give informed consent
* English-speaking

Exclusion Criteria:

* Patients experiencing tinnitus related to cochlear implantation, retrocochlear lesion, or other known anatomic/structural lesions of the ear and temporal bone
* Patients with hyperacusis or misophonia (hyper-sensitivity to loud noises)
* Patients with cardiac pacemakers, intracardiac lines, implanted medication pumps, implanted electrodes in the brain, other intracranial metal objects with the exception of dental fillings, or any other contraindication for MRI scan
* Patients with an acute or chronic unstable medical condition which, in the opinion of the investigator, would require stabilization prior to initiation of magnetic stimulation
* Patients with any active ear disease that, in the opinion of the PI, needs to be further evaluated
* Patients with symptoms of depression as evidenced by a score of 14 or greater on the Beck Depression Inventory or, in the opinion of the psychiatric sub-investigator demonstrates active mood symptoms that meet DSM-IV-TR criteria for Major Depressive Disorder
* Any psychiatric co-morbidity that, in the opinion of the psychiatric sub-investigator, may complicate the interpretation of study results
* Patients with tinnitus related to Workman's Compensation claim or litigation-related event
* Weight over 350 pounds
* A Mini-Mental Status Exam score less than 27
* Patients with a history of claustrophobia
* Inability to lay flat for 2 hours
* Active alcohol and/or drug dependence or history of alcohol and/or drug dependence within the last year
* Any medical condition that, in the opinion of the investigators, confounds study results or places the subject at greater risk
* Unable to provide informed consent
* Any exclusions from radiology screening Currently Pregnant

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 19 adults between the ages of 45 and 60 years, age and hearing level-matched to the bothered tinnitus cohort from the on-going research at Washington University. Subjects will be recruited from an institutional tinnitus database, from Washington University Otolaryngology Clinics, as well as the general public through poster advertisement on the Washington University grounds.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre M Wineland, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, Center for Clinical Studies, St Louis, Missouri, United States

REFERENCES:
- [Result] Wineland AM, Burton H, Piccirillo J. Functional connectivity networks in nonbothersome tinnitus. Otolaryngol Head Neck Surg. 2012 Nov;147(5):900-6. doi: 10.1177/0194599812451414. Epub 2012 Jun 21. PMID 22722065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Those with subjective, idiopathic tinnitus were recruited from WU audiology and otolaryngology clinics.
Pre-assignment Details: 1 participant was excluded due to claustrophobia from the MRI and another participant withdrew midway through the neurocognitive evaluation due to frustration.
Groups:
- Non-Bothered Tinnitus Group: Participants who answer no bother or slight bother on a global tinnitus bothersome score. Tinnitus Handicap Index <30.
Period: Overall Study
Arm/Group | Non-Bothered Tinnitus Group
Started | 20
Completed | 18
Not Completed | 2
Not completed — Claustrophibia and Frustration | 2

BASELINE CHARACTERISTICS:
Arm/Group | Non-Bothered Tinnitus Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in Blood Oxygen Level as Measured by Functional Connectivity MRI
Description: Perform Functional connectivity MRI on participants with non-bothersome tinnitus. By undergoing a functional MRI, we are able to delineate the various networks involved with tinnitus including the default mode, attention, auditory, visual, somatosensory, and cognitive networks. The functional connectivity differences are measured by changes in blood oxygen level changes.
Time Frame: 8 months for complete analysis on all participants
Population: Perform Functional Connectivity MRI on Participants With Non-bothersome Tinnitus. Non-Bothered Tinnitus Group includes participants who answer 'no bother' or 'slight bother' on a global tinnitus bothersome scale and less than 30 on the Tinnitus Handicap Index.
Measure: Number; unit: participants
Groups:
- Non-Bothered Tinnitus Group: Perform Functional Connectivity MRI on Participants With Non-bothersome Tinnitus. Participants who answer no bother or slight bother on a global tinnitus bothersome score. Tinnitus Handicap Index <30.
Arm/Group | Non-Bothered Tinnitus Group
Number analyzed (Participants) | 18
participants | 18
Statistical Analysis 1: Comparison: Non-Bothered Tinnitus Group; Null hypothesis: Fisher's transform z scores for a seed region were comparable between the control and non-bothered tinnitus groups; Test type: Other — The analysis is based on a threshold-free cluster enhancement permutation technique; p < 0.01, Fisher Exact — all correlations were transformed into z scores using Fisher's transformation and a t test evaluated group differences; The analysis is based on a threshold-free cluster enhancement permutation technique

ADVERSE EVENTS:
Arm/Group | Non-Bothered Tinnitus Group
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No